CLINICAL TRIAL: NCT05590832
Title: The Effect of Smart-Phone Interventional Messages on Gestational Weight Gain: A Randomized Controlled Study
Brief Title: The Effect of Smart-Phone Interventional Messages on Gestational Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Yıldız, Research Assistant Gizem Yıldız (Master Student), Ordu University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Gy1995
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gestational Weight Gain
Keywords: pregnancy; gestational weight gain; weight gain during pregnancy; healthy eating; physical exercise
MeSH Terms: conditions — Gestational Weight Gain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The individuals included in the study were first stratified according to their BMI classes (normal, preobese, obese). Then, the BMI classes were included in the experimental and control groups in a balanced way by block randomisation method. Within each stratum, randomisation lists were generated with the help of "The random sorting randomization algorithm" (Maximum Allowable Deviation = 10%) PASS 11.0 software (NCSS LLC, Kaysville, UT). In total, participants were randomly assigned to experimental and control groups of 51 participants each.The study was completed with 96 pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İnitiative group (Experimental): All pregnant women participating in the study were divided into intervention and control groups by applying randomization. Pre-test data of both groups will be collected before 18th gestational week, and post-test data will be collected after 37th gestational week.
  Pregnant women assigned to the initiative group were added to a group established via Whatsapp. Information messages will be sent via Whatsapp on Mondays, Wednesdays and Fridays for the first 10 weeks / three times a week (up to the 28th week), and reminder messages will be sent once a week on Wednesdays between the 29th-36th weeks. When necessary, individual messages will be sent to the pregnant women and special directions will be given according to their weight gain rates.
  Interventions: Behavioral: Activity of Whatsapp messages
- Control group (No Intervention): In the same way, a Whatsapp group will be set up to the control group and messages will be sent once a month about the subjects included in antenatal care up to 37 weeks. Topics included in routine maintenance will be included.

INTERVENTIONS:
Behavioral: Activity of Whatsapp messages — Informative messages will be sent to the initiative group on Mondays, Wednesdays and Fridays for the first 10 weeks / three times a week (up to the 28th week), and reminder messages will be sent once a week on Wednesdays between the 29th-36th weeks.
  Arms: İnitiative group

SUMMARY:
Methods: The study is a randomized controlled experimental study. Groups were determined by stratified randomization according to the BMI of the pregnant women. In the study, individual identification form, Healthy Living Behaviors in Pregnancy Scale (HLBPS), and maternal questionnaire were used. The initiative program was carried out via WhatsApp messages on a smartphone. Messages regarding routine prenatal care were sent to the intervention group three times a week, and to the control group once a month, about appropriate weight gain, nutrition, and physical activity via WhatsApp.

Results: The mean gestational weight gain was 13.1±4.3 in the intervention group and 14.6±4.2 in the control group, and no significant difference was found between the groups. According to the IOM guideline, there was a significant difference between the groups in terms of appropriate GWG , while no significant difference was found between excessive GWG.HLBPS scale total score, nutrition and physical activity post-test mean scores increased significantly in the intervention group compared to the control group. In the intervention group, the group/time interaction in the scale total score, nutrition and physical activity scores of the pregnant women who gained appropriate weight according to the IOM guideline was significant, and the intervention was effective.Significant differences were found between the groups in the pretest-posttest score differences in the HLBPS total score, nutrition and physical activity sub-dimensions of the pregnant women.

Conclusion: Healthy nutrition and physical activity short message intervention with a smart phone increased the appropriate gestational weight gain rates of pregnants in the intervention group according to the IOM guideline, and the intervention was effective. However, there was no difference between the groups in terms of excessive gestational weight gain. It is recommended to conduct studies with a high level of evidence, including internet and social media applications, with larger samples.

DETAILED DESCRIPTION:
Most of the descriptive characteristics of the intervention and control group pregnant women who participated in the study were homogenously distributed (p>0.05). A significant difference was found only between gestational week and place of residence (p<0.05).The mean total GWG of all pregnant women participating in the study was 13.9±4.3/kg. The mean difference between the intervention (13.1±4.3/kg) and control group (14.6±4.2/kg) pregnant women was 1.5 kg, but no significant difference was found between the groups (p>0.05). The rate of GWG within the limits of IOM guideline recommendations in the intervention group pregnant women (48.9%) was significantly higher than in the control group (22.2%) (p<0.05). Excessive GWG was found to be higher in the control group (68.9%) than in the intervention group (48.9%), but no significant difference was found (p>0.05).In the pre-intervention, pre-test data, pregnancy responsibility, nutrition and physical activity and HLBPS total scores were higher in the intervention group than in the control group (p<0.05). While no significant difference was found between the groups in the post-test scores of the pregnancy responsibility sub-dimension of the intervention/control group pregnant women (p>0.05), a statistically significant difference was found in both intervention (p<0.001) and control groups (p<0.001) in the in-group pre-post comparison. While there was a significant increase in the intra-group nutrition, physical activity sub-dimension and HLBPS total score of the intervention group pregnant women (p<0.001), no significant increase was observed in the control group (p>0.05). In the post-test comparison between groups, nutrition, physical activity sub-dimension score and HLBPS total score increased significantly in the intervention group compared to the control group (p<0.001). While the nutrition sub-dimension score of the intervention group was effective in appropriate GWG, it was not effective in the control group. Physical activity sub-dimension and HLBPS total score were effective in appropriate GWG in both intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18-45,

* Using Whatsapp,
* Having a smart phone and using the internet,
* At least primary school graduate/literate,
* Does not have any chronic and psychological disorders,
* Having spontaneous pregnancy,
* Volunteer to participate in the research,
* Pregnancy below the 16th week of participation in the study,
* Not having any physical disability,
* Pregnant women with low pregnancies with low BMI and not morbidly obese were included in the study.

Exclusion Criteria:

Dropping out of research participation and initiative program,

* Low,
* Giving birth before 37 weeks,
* Having multiple pregnancy,
* Those who did not have a spontaneous pregnancy were not included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is a study conducted with pregnant women.
Enrollment: 96 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Gestational Weight Gain | Total amount of weight gained until 37 weeks of pregnancy
  Gestational weight gain rate in line with IOM guideline, Thanks to the intervention, it is expected that the average weight gain of the pregnant women in the intervention group will be lower than the control group.
Appropriate GWG ratios with IOM guideline | Compliance status of the total weight gained until the 37th week of pregnancy according to the IOM guideline
  Compliance with the IOM guideline 2009,Thanks to the intervention, it is expected that the pregnant women in the intervention group will have higher rates of appropriate weight gain according to the 2009 IOM guideline compared to the control group.
Healthy living behavior scale score | at the end of 37th week of pregnancy
  healthy living behavior scale score in pregnant women

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No